CLINICAL TRIAL: NCT02541773
Title: The Characterisation of Vascular Biomarkers Before and After Cardiac Resynchronization Therapy in Patients With Chronic Heart Failure and Their Role in Predicting Response
Brief Title: Novel Vascular Biomarkers Behaviour and Clinical Value in Heart Failure and CRT
Acronym: COVERT-HF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr Christopher McAloon, Cardiology Research Fellow, University Hospitals Coventry and Warwickshire NHS Trust
Other Study IDs: version 10 20 Jan 2016
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Cardiac Resynchronization Therapy; Vascular Biomarker; miRNA; Extracellular Matrix; Brain Natruetic Peptide; Growth Degradation Factor-15; Body Composition
MeSH Terms: interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants with have peripheral and coronary sinus samples taken for plasma and serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Heart Failure Patients: Undergoing CRT implantation, all will be observed for 6 months and will be defined at the end of the observation period as responder or non-responder
  Interventions: Device: Cardiac Resynchronisation Therapy

INTERVENTIONS:
Device: Cardiac Resynchronisation Therapy — Routine implantation of CRT - part of standard of care

SUMMARY:
The purpose of this study is to understand the behaviour of certain blood markers in patients with heart failure who undergo a cardiac device implantation procedure called cardiac resynchronization therapy (CRT). CRT is an effective treatment for heart failure, but up to 30% of people do not respond and have poor outcomes (1,2). Despite extensive investigation, identifying these patients continues to be a challenge. The study intends to describe the changes in these blood markers before and after CRT and to examine any potential clinical value.

The idea behind the study is that these blood markers alter in heart failure and change with CRT implantation. Furthermore the pattern of marker expression before implant and after may predict response and outcome.

DETAILED DESCRIPTION:
Study Design A prospective, non-randomised, self-control study of unselected heart failure patients undergoing CRT implantation, all recruited within two years All participants having CRT implantation at University Hospital Coventry and Warwickshire will be screened using the eligibility criteria (outlined below).

Participants will have three assessments within six months (baseline, 6 weeks and 6 months approximately). All visits coincide with routine clinical visits for CRT implantation and interrogation. Assessments at all three time points will include clinical data (including New York Heart Association functional class), quality of life measurements (Minnesota Living with Heart Failure questionnaire), echocardiography data (left ventricular volumetric assessment, ejection fraction), electrocardiograph, functional capacity (6 minute-walk test) and body composition assessment (air displacement). Peripheral blood samples will be taken to examine novel vascular biomarkers and to examine renal function, full blood count, diabetic control (HBA1c - only diabetics) and Brain Natruetic Peptide. Coronary sinus samples will be taken for novel vascular biomarkers in a small proportion of the cohort.

Blood Sampling and Storage

Participants are asked to starve for two hours and rest for one hour before blood sampling. Coronary sinus blood sampling occurs at the time of coronary sinus cannulation before contrast is injected. Blood samples (serum/plasma) are taken in citrate and EDTA tubes. The samples stand at room temperature for a minimum of 30 minutes and undergo centrifugation within an hour. Centrifugation (3500rpm for 10 minutes) occurs at room temperature. Samples are then stored in -80 freezer.

Laboratory Analysis

Samples will undergo final analysis at the University of Warwick and Kings College London. Novel vascular biomarkers of heart failure that exist as proteins in the serum will be analysed using enzyme-linked immunosorbent assay (ELISA) techniques previously outlined in publications (3-6). The specific novel vascular biomarkers represent different aspects of adverse ventricular remodelling; myocardial stress [Growth Differentiation Factor-15] and extracellular remodelling [Matrix Metalloproteinases -2 & -9, Aminoterminal Propeptides of Type I Collagen (PINP), Aminoterminal Propeptides of Type III Collagen (PIIINP), Carboxy-Terminal Telopeptide of Type I Collagen (CITP)] (4-7). These markers will undergo quantification using ELISA techniques that have previously described in the literature (8, 9).

Micro Ribonucleic Acids (miRNA) profiling will be undertaken in coronary sinus and peripheral samples and will be compared to those taken after CRT implantation. Responders will be compared to non-responders to determine variation in profile between these two distinct groups. Profiling and quantification will be performed as described in previous publications (10-12). Specific cardiac miRNA will be pre-selected to screen and quantify, especially those have already been proven to have altered expression in heart failure (13-16).

Device Implantation

CRT devices (pacemaker of defibrillator) are implanted by two independent operators at our single centre in a standard fashion. CRT is implanted traditionally in the left deltopectoral groove. Venous access is via the cephalic>axillary>subclavian veins (all operators can cannulate either vein based on individual patient). Right ventricular lead for the majority of patients will be implanted at the right ventricular apex. Right atrial leads will be planned to be implanted in the right atrial appendage. Patients in permanent Atrial Fibrillation will not have a right atrial lead implanted. Coronary sinus will be cannulated and angiography performed to roadmap anatomy for lead deployment site. The most lateral position will be favoured in a basal/ mid-cavity position. At the point of coronary sinus cannulation blood samples (plasma/serum will be taken). Post procedure patients undergo targeted echocardiography and a chest x-ray film. Post procedure on the day of implant patients will undergo CRT interrogation and optimisation of programming.

Echocardiography

A focused echocardiographic study assessing the left ventricle will be performed to the recommended international standard (17). The left ventricular systolic and diastolic function will be fully assessed. Volumetric assessment will be performed using Simpson's method (17). Diastolic function will be assessed by performing volumetric assessment of the left atrium, measuring pulse wave inflow of ventricular filling and TDI of the lateral and septal walls [apical 4 chamber]. All scans will be performed on the departmental machines [GE systems, Vivid 7] and by the same operator. Scans will be performed independently and previous scans will not have been reviewed before this scan. Full analysis will be conducted once all scans have been performed.

Inter- and Intra-Observer Variability Echocardiography Study

An inter- and intra-observer variability study will be performed to ensure standardisation of echocardiographic examinations. Twenty percent of echocardiograms will be randomly selected to have measurements and conclusions reviewed. An independent cardiologist/ cardiac physiologist (accredited by the British Society of Echocardiography) will be blinded to selected echocardiograms and will validate reporting and measurements of these examinations.

Body Composition

Air-displacement plethysmography (Bodpod) is an easily accessible and safe tool to measure body composition (18). The assessment is reproducible and is comparable to other measures of body composition (18). The major advantage of Bodpod is that it is safe for patients who have had a CRT implanted. The University of Warwick and University Hospital Coventry and Warwickshire (UHCW) has one of the few facilities in their Human Metabolic Unit to perform Bodpod.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Left ventricular ejection fraction ≤35% on echocardiography
3. NYHA Class III/IV symptoms or milder symptoms with:

   * NYHA I (LVEF <35% and QRS>150msec on resting ECG)
   * NYHA II (LVEF <35% with either QRS>150msec or QRS 120-149msec with Left Bundle Branch Block on resting ECG)
4. Optimal medical therapy for heart failure that the patient tolerates (ACEi, Beta-Blocker, Mineralocorticoid) for > 3 months
5. QRS duration ≥120-149msec with LBBB on resting ECG or QRS duration >150msec on resting ECG
6. Patient consent to participation in the study

Exclusion Criteria:

1. Acute heart failure decompensation < 6/52 before implant
2. Significant cognitive impairment
3. Acute coronary syndrome < 6/52 before implant
4. Chronic kidney disease stage V (requiring dialysis)
5. Terminal illness with likely survival < 1 year after implant

Post Procedure Exclusions:

1. Failure of procedure (e.g. coronary sinus anatomy) 2. Complication resulting in poor/ none biventricular pacing (e.g. phrenic nerve stimulation, lead displacement/ damage)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic heart failure patients who have been referred for and meet national criteria for Cardiac Resynchronization Therapy implants
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Response | 6 months
  Two of three criteria must be fulfilled to be defined as a clinical response:
  1. New York Heart Association (NYHA) > 1 class reduction from baseline
  2. Minnesota Living with Heart Failure Questionnaire (MLHFQ) score < 5 from baseline
  3. Six minute walk test (6MWT) increase in baseline distance by 10%
  Mortality or heart transplantation within 6 months of implant will be defined as a non-response.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular Outcomes | 12 months
  Composite score of all-cause mortality and first heart failure hospitalisation (admission requiring intravenous diuretics)
Echocardiographic Response | 6 months
  ≥15% reduction in left ventricular end-systolic volume

CONTACTS AND LOCATIONS:
Overall Officials: Faizel Osman, MD FRCP FESC, Principal Investigator — University Hospital Coventry and Warwickshire
Locations (1):
- University Hospital Coventry and Warwickshire, Coventry, Warwickshire, United Kingdom

REFERENCES:
- [Background] Cleland JG, Daubert JC, Erdmann E, Freemantle N, Gras D, Kappenberger L, Tavazzi L; Cardiac Resynchronization-Heart Failure (CARE-HF) Study Investigators. The effect of cardiac resynchronization on morbidity and mortality in heart failure. N Engl J Med. 2005 Apr 14;352(15):1539-49. doi: 10.1056/NEJMoa050496. Epub 2005 Mar 7. PMID 15753115
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Garcia-Bolao I, Macias A, Lopez B, Gonzalez A, Gavira JJ, Azcarate P, Alegria E, Diez J. A biomarker of myocardial fibrosis predicts long-term response to cardiac resynchronization therapy. J Am Coll Cardiol. 2006 Jun 6;47(11):2335-7. doi: 10.1016/j.jacc.2006.03.012. Epub 2006 May 16. No abstract available. PMID 16750706
- [Background] Garcia-Bolao I, Lopez B, Macias A, Gavira JJ, Azcarate P, Diez J. Impact of collagen type I turnover on the long-term response to cardiac resynchronization therapy. Eur Heart J. 2008 Apr;29(7):898-906. doi: 10.1093/eurheartj/ehn098. Epub 2008 Mar 10. PMID 18334474
- [Background] Hessel MH, Bleeker GB, Bax JJ, Henneman MM, den Adel B, Klok M, Schalij MJ, Atsma DE, van der Laarse A. Reverse ventricular remodelling after cardiac resynchronization therapy is associated with a reduction in serum tenascin-C and plasma matrix metalloproteinase-9 levels. Eur J Heart Fail. 2007 Oct;9(10):1058-63. doi: 10.1016/j.ejheart.2007.07.007. Epub 2007 Aug 28. PMID 17728181
- [Background] Umar S, Bax JJ, Klok M, van Bommel RJ, Hessel MH, den Adel B, Bleeker GB, Henneman MM, Atsma DE, van der Wall EE, Schalij MJ, van der Laarse A. Myocardial collagen metabolism in failing hearts before and during cardiac resynchronization therapy. Eur J Heart Fail. 2008 Sep;10(9):878-83. doi: 10.1016/j.ejheart.2008.06.019. Epub 2008 Sep 2. PMID 18768351
- [Background] Foley PW, Stegemann B, Ng K, Ramachandran S, Proudler A, Frenneaux MP, Ng LL, Leyva F. Growth differentiation factor-15 predicts mortality and morbidity after cardiac resynchronization therapy. Eur Heart J. 2009 Nov;30(22):2749-57. doi: 10.1093/eurheartj/ehp300. Epub 2009 Aug 7. PMID 19666898
- [Background] Lewandowski KC, Komorowski J, Mikhalidis DP, Bienkiewicz M, Tan BK, O'Callaghan CJ, Lewinski A, Prelevic G, Randeva HS. Effects of hormone replacement therapy type and route of administration on plasma matrix metalloproteinases and their tissue inhibitors in postmenopausal women. J Clin Endocrinol Metab. 2006 Aug;91(8):3123-30. doi: 10.1210/jc.2005-2789. Epub 2006 May 16. PMID 16705077
- [Background] Randeva HS, Lewandowski KC, Komorowski J, Murray RD, O'Callaghan CJ, Hillhouse EW, Stepien H, Shalet SM. Growth hormone replacement decreases plasma levels of matrix metalloproteinases (2 and 9) and vascular endothelial growth factor in growth hormone-deficient individuals. Circulation. 2004 May 25;109(20):2405-10. doi: 10.1161/01.CIR.0000129763.51060.77. Epub 2004 May 3. PMID 15123527
- [Background] Zampetaki A, Kiechl S, Drozdov I, Willeit P, Mayr U, Prokopi M, Mayr A, Weger S, Oberhollenzer F, Bonora E, Shah A, Willeit J, Mayr M. Plasma microRNA profiling reveals loss of endothelial miR-126 and other microRNAs in type 2 diabetes. Circ Res. 2010 Sep 17;107(6):810-7. doi: 10.1161/CIRCRESAHA.110.226357. Epub 2010 Jul 22. PMID 20651284
- [Background] Willeit P, Zampetaki A, Dudek K, Kaudewitz D, King A, Kirkby NS, Crosby-Nwaobi R, Prokopi M, Drozdov I, Langley SR, Sivaprasad S, Markus HS, Mitchell JA, Warner TD, Kiechl S, Mayr M. Circulating microRNAs as novel biomarkers for platelet activation. Circ Res. 2013 Feb 15;112(4):595-600. doi: 10.1161/CIRCRESAHA.111.300539. Epub 2013 Jan 2. PMID 23283721
- [Background] Zampetaki A, Mayr M. Analytical challenges and technical limitations in assessing circulating miRNAs. Thromb Haemost. 2012 Oct;108(4):592-8. doi: 10.1160/TH12-02-0097. Epub 2012 May 25. PMID 22627831
- [Background] Romaine SP, Tomaszewski M, Condorelli G, Samani NJ. MicroRNAs in cardiovascular disease: an introduction for clinicians. Heart. 2015 Jun;101(12):921-8. doi: 10.1136/heartjnl-2013-305402. Epub 2015 Mar 26. PMID 25814653
- [Background] Marfella R, Di Filippo C, Potenza N, Sardu C, Rizzo MR, Siniscalchi M, Musacchio E, Barbieri M, Mauro C, Mosca N, Solimene F, Mottola MT, Russo A, Rossi F, Paolisso G, D'Amico M. Circulating microRNA changes in heart failure patients treated with cardiac resynchronization therapy: responders vs. non-responders. Eur J Heart Fail. 2013 Nov;15(11):1277-88. doi: 10.1093/eurjhf/hft088. Epub 2013 Jun 4. PMID 23736534
- [Background] Vogel B, Keller A, Frese KS, Leidinger P, Sedaghat-Hamedani F, Kayvanpour E, Kloos W, Backe C, Thanaraj A, Brefort T, Beier M, Hardt S, Meese E, Katus HA, Meder B. Multivariate miRNA signatures as biomarkers for non-ischaemic systolic heart failure. Eur Heart J. 2013 Sep;34(36):2812-22. doi: 10.1093/eurheartj/eht256. Epub 2013 Jul 17. PMID 23864135
- [Background] Tijsen AJ, Creemers EE, Moerland PD, de Windt LJ, van der Wal AC, Kok WE, Pinto YM. MiR423-5p as a circulating biomarker for heart failure. Circ Res. 2010 Apr 2;106(6):1035-9. doi: 10.1161/CIRCRESAHA.110.218297. Epub 2010 Feb 25. PMID 20185794
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Fields DA, Goran MI, McCrory MA. Body-composition assessment via air-displacement plethysmography in adults and children: a review. Am J Clin Nutr. 2002 Mar;75(3):453-67. doi: 10.1093/ajcn/75.3.453. PMID 11864850
- [Derived] McAloon CJ, Barwari T, Hu J, Hamborg T, Nevill A, Hyndman S, Ansell V, Musa A, Jones J, Goodby J, Banerjee P, O'Hare P, Mayr M, Randeva H, Osman F. Characterisation of circulating biomarkers before and after cardiac resynchronisation therapy and their role in predicting CRT response: the COVERT-HF study. Open Heart. 2018 Oct 18;5(2):e000899. doi: 10.1136/openhrt-2018-000899. eCollection 2018. PMID 30364565